CLINICAL TRIAL: NCT03072797
Title: Beijing Hospital Atherosclerosis Study
Acronym: BHAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Fusui Ji, MD, Director, Department of Gerontological Cardiology, Beijing Hospital
Other Study IDs: 2016BJYYEC-121-02
Record Dates: First submitted 2017-02-27; First posted 2017-03-07 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Stroke
Keywords: Atherosclerosis; Longitudinal; Biomarker; Coronary angiography; Follow-up; Metabolomics; Risk factor
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, 10 mL (whole blood, plasma, serum)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Beijing Hospital Atherosclerosis Study (BHAS) is a prospective, single-center, observational cohort study performed at the Beijing Hospital in Beijing, China. Subjects enrolled in this study will be the consecutive patients undergoing coronary angiography in the hospital. Blood samples are taken immediately before the angiographic procedure. Clinical and angiographic characteristics are recorded. All patients will have routine follow-up at 6 months and 1 year postprocedure, then yearly thereafter. Follow-up includes mortality, myocardial infarction (MI), stroke, rehospitalization, coronary revascularization procedures, life styles, and medication use. The primary end point for the study will be the major adverse cardiovascular events (MACE), defined as death from any cause, nonfatal myocardial infarction, nonfatal stroke and revascularization. This study has been reviewed and approved by the Ethics Committee of Beijing Hospital. All enrolled individuals will be received written notice of the intended use of their blood samples and provided written consent.

The major objectives of the BHAS Study are to (1) establish a prospective cohort and a biological sample bank in ethnic Chinese with coronary angiography, (2) identify baseline new biosignature profiles such as novel biomarkers via metabolomics approach associated with the subsequent clinical events, (3) assess the use of molecular profiles from multiple platforms (eg, genomics, proteomics, and metabolomics) integrated with readily available clinical information for improved risk classification for cardiovascular events, and (4) provide clearer understanding of underlying disease processes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18y
* Consent for the study
* Primary reason for catheterization is concern for ischemic heart disease
* Complete clinical and coronary angiogram data available

Exclusion Criteria:

* Primary pulmonary hypertension or severe lung disease
* Cardiac transplantation
* Other solid organ transplant
* Peripheral vascular intervention only
* Right heart catheterization only
* Advanced heart failure
* Congenital heart disease
* Women who are pregnant or nursing, or preparing for pregnant during the study period
* Progressive fatal disease
* History of alcoholism or drug abuse
* Patients with mental illness and are being treated
* Patients are undergoing radiotherapy or chemotherapy
* Acute and chronic infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in this study will be the consecutive patients undergoing coronary angiography at the Beijing Hospital in Beijing, China.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major adverse cardiovascular events (MACE) | 3 years
  MACE include death from any cause, nonfatal myocardial infarction, nonfatal stroke and revascularization.

SECONDARY OUTCOMES:
Number of participants with other atherosclerosis events | 3 years
  Other atherosclerosis events include readmission for angin and transient ischemic attack.

CONTACTS AND LOCATIONS:
Overall Officials: Fusui Ji, M.D., Principal Investigator — Department of Cardiology, Beijing Hospital,National Center of Gerontology; Wenxiang Chen, M.D., Principal Investigator — The MOH Key Laboratory of Geriatrics, Beijing Hospital, National Center of Gerontology; Xue Yu, M.D., Principal Investigator — Department of Cardiology, Beijing Hospital,National Center of Gerontology
Locations (1):
- Bejing Hosptial, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Kip KE, Hollabaugh K, Marroquin OC, Williams DO. The problem with composite end points in cardiovascular studies: the story of major adverse cardiac events and percutaneous coronary intervention. J Am Coll Cardiol. 2008 Feb 19;51(7):701-7. doi: 10.1016/j.jacc.2007.10.034. PMID 18279733
- [Background] Ussher JR, Elmariah S, Gerszten RE, Dyck JR. The Emerging Role of Metabolomics in the Diagnosis and Prognosis of Cardiovascular Disease. J Am Coll Cardiol. 2016 Dec 27;68(25):2850-2870. doi: 10.1016/j.jacc.2016.09.972. PMID 28007146
- [Derived] Wang Y, Yang R, Zhang Y, Wang Z, Wang X, Wang S, Zhang W, Yu X, Dong J, Chen W, Ji F. Prognostic Value of Serum 1,5-anhydroglucitol Levels in Patients with Acute Myocardial Infarction. Rev Cardiovasc Med. 2022 Dec 2;23(12):394. doi: 10.31083/j.rcm2312394. eCollection 2022 Dec. PMID 39076658
- [Derived] Yang R, Zhang W, Wang X, Wang S, Zhou Q, Li H, Mu H, Yu X, Ji F, Dong J, Chen W. Nonlinear association of 1,5-anhydroglucitol with the prevalence and severity of coronary artery disease in chinese patients undergoing coronary angiography. Front Endocrinol (Lausanne). 2022 Sep 5;13:978520. doi: 10.3389/fendo.2022.978520. eCollection 2022. PMID 36133308